CLINICAL TRIAL: NCT03671343
Title: Impact of Physical Rehabilitation on Sarcopenia Inolder and Chronic Kidney Patients
Brief Title: Physical Rehabilitation and Chronic Kidney Disease
Acronym: IMPREPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL17_0598
Record Dates: First submitted 2017-10-10; First posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Sarcopenia; Chronic Kidney Disease; Older
Keywords: sarcopenia; chronic kidney disease; older
MeSH Terms: conditions — Sarcopenia; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention : Physical rehabilitation (Experimental): The Arm "Physical rehabilitation" will benefit from the implementation of the "Loss of Mobility Prevention" program set up in the Department of Aging Medicine of the Center Hospitalier Lyon Sud (CHLS) of Pr BONNEFOY.
  Interventions: Behavioral: Physical rehabilitation
- Control : optimized medical treatment (No Intervention): The Arm "Optimized medical treatment" will not benefit from the implementation of the "Loss of Mobility Prevention" program.

INTERVENTIONS:
Behavioral: Physical rehabilitation — It will benefit from an initial and final geriatric assessment, an initial dietary balance and a personalized treatment in physical activities adapted for 3 months by an Educator in Adapted Physical Activities.
  Arms: Intervention : Physical rehabilitation

SUMMARY:
Older patients with chronic renal failure suffer from sarcopenia. Loss of muscle function is associated with increased morbidity and mortality. Currently few treatment are available. The aim of this study is to evaluate the impact of physical rehabilitation in this population on muscle performance and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* man or woman
* age over 70 years
* CKD stage 3B, 4 or 5 or a DFG <45ml / min according to CKD-EPI formula
* an SPPB (Short Physical Performance Battery test )<10
* having received a complete and loyal information and having given his written and informed consent.
* ability to rehabilitate

Exclusion Criteria:

* Subject not presenting previous inclusion criteria
* General condition not compatible for the realization of physical rehabilitation
* Patient protected under the terms of the law.
* Inability to respect the follow-up of the study for geographical, social or psychological reasons.
* depression or other psychiatric disorder
* Refusal to participate in the study
* Absence of affiliation to the social security system
* Subject in a exclusion period of an other study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline distance travelled (in meters) during the 6-minute walking distance (6MWD) test (muscular performance), at 3 months | Baseline and 3 months

SECONDARY OUTCOMES:
Nutritional parameter: Albuminemia | Baseline,3 and 6 months
Nutritional parameter: Prealbuminemia | Baseline,3 and 6 months
Nutritional parameter: Body mass index | Baseline,3 and 6 months
Nutritional parameter: bioimpedancemetry | Baseline,3 and 6 months
Muscle strength evaluated by Hand Grip strength test | Baseline,3 and 6 months
Quality of life evaluated by the questionnaire SF-36 (36-item medical outcomes study Short-Form health survey) | Baseline,3 and 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service de Médecine du vieillissement, soins de suite et de rééducation, Centre Hospitalier Lyon SUd, Pierre-Bénite
  - Service de Néphrologie, Centre Hospitalier Lyon Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No